CLINICAL TRIAL: NCT05940415
Title: Conducting Active Surveillance Without Prostate Biopsy for Patients With Low-risk Suspected Prostate Cancer Based on USTC Diagnostic Model and PSA Level: a Multicenter Prospective Study
Brief Title: Conducting Active Surveillance Without Prostate Biopsy for Patients With Low-risk Suspected Prostate Cancer
Acronym: ASWBP
Status: Recruiting | Type: Observational
Sponsor: Anhui Provincial Hospital (Other Government)
Collaborators: Zhongda Hospital (Other); Wannan Medical College Yijishan Hospital (Other); Wuhu City Second People's Hospital (Other)
Responsible Party: Principal Investigator, TaoTao, Associate professor, Associate chief physician, Anhui Provincial Hospital
Other Study IDs: SNOTOB-II
Record Dates: First submitted 2023-06-28; First posted 2023-07-11 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; prostate biospy; mpMRI; prostate specific antigen density; diagnostic model; active surveillance
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with low-risk of prostate cancer based on USTC diagnostic model and serum PSA levels.: Patients with PSA between 4 to 10 ng/ml and USTC model predicted probability of cancer less than 0.05 (https://ustcprostatecancerprediction.shinyapps.io/dynnomapp/).
  Interventions: Behavioral: active surveillance

INTERVENTIONS:
Behavioral: active surveillance — active surveillance without prostate biopsy

SUMMARY:
The goal of this observational study is to evaluate the role of the USTC diagnostic model in risk-adaptive strategies for biopsy decision-making in patients with low-risk suspected prostate cancer in order to reduce unnecessary biopsy. Based on the USTC diagnostic model (website: https://ustcprostatecancerprediction.shinyapps.io/dynnomapp/) and serum PSA levels, patients with low-risk suspected prostate cancer are enrolled and received active surveillance rather than biopsy. The main questions to be answered is:

• The safety and feasibility of conducting biopsy-free active monitoring in patients with low-risk suspected prostate cancer accessed by the USTC diagnostic model and serum PSA levels.

Participants will be required to undergo serum PSA testing every 3 months, mpMRI testing every 6 months, and reassessment of the probability of developing prostate cancer using the USTC model every 3 months. Patients who do not meet the inclusion criteria and are at increased risk will no longer receive active surveillance and will be advised to undergo biopsy. Dynamic changes in PI-RADS score and biopsy results will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with clinically suspected PCa have indications for prostate biopsy;
2. Complete serum PSA testing and mpMRI examination in the outpatient department;
3. 4 ng/ml ≤ serum total PSA ≤10 ng/ml;
4. The probability of prostate cancer calculated by USTC diagnostic models is less than 0.05;
5. There is no family history of prostate cancer and no history of other malignant tumors.

Exclusion Criteria:

1. The patient has previous history of prostate biopsy;
2. Lack of complete clinical information, such as failure to perform mpMRI;
3. Patients with serum total PSA < 4ng/ml or > 10ng/ml.
4. According to USTC diagnostic model, the probability of prostate cancer is equal or more than 0.05.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We select patients with low-risk suspected prostate cancer evaluated by USTC diagnostic model and serum PSA level. After meeting the inclusion criteria, follow-up surveys will be conducted.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2023-10-08 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
prostate cancer diagnostic free survival time | through study completion, an average of 2 year
  survival analysis by K-M curves and log-rank tests

SECONDARY OUTCOMES:
dynamic change of serum total PSA | every 3 months up to 2 years
  dynamic change serum PSA level after active surveillance
dynamic change of PI-RADS score | every 6 months up to 2 years
  dynamic change PI-RADS score after active surveillance

CONTACTS AND LOCATIONS:
Overall Officials: Tao Tao, Study Chair — The First Affiliated Hospital of USTC
Locations (1):
- The First Affiliated Hospital of USTC, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xia C, Dong X, Li H, Cao M, Sun D, He S, Yang F, Yan X, Zhang S, Li N, Chen W. Cancer statistics in China and United States, 2022: profiles, trends, and determinants. Chin Med J (Engl). 2022 Feb 9;135(5):584-590. doi: 10.1097/CM9.0000000000002108. PMID 35143424
- [Background] Ilic D, Djulbegovic M, Jung JH, Hwang EC, Zhou Q, Cleves A, Agoritsas T, Dahm P. Prostate cancer screening with prostate-specific antigen (PSA) test: a systematic review and meta-analysis. BMJ. 2018 Sep 5;362:k3519. doi: 10.1136/bmj.k3519. PMID 30185521
- [Background] Mottet N, van den Bergh RCN, Briers E, Van den Broeck T, Cumberbatch MG, De Santis M, Fanti S, Fossati N, Gandaglia G, Gillessen S, Grivas N, Grummet J, Henry AM, van der Kwast TH, Lam TB, Lardas M, Liew M, Mason MD, Moris L, Oprea-Lager DE, van der Poel HG, Rouviere O, Schoots IG, Tilki D, Wiegel T, Willemse PM, Cornford P. EAU-EANM-ESTRO-ESUR-SIOG Guidelines on Prostate Cancer-2020 Update. Part 1: Screening, Diagnosis, and Local Treatment with Curative Intent. Eur Urol. 2021 Feb;79(2):243-262. doi: 10.1016/j.eururo.2020.09.042. Epub 2020 Nov 7. PMID 33172724
- [Background] Duffy MJ. Biomarkers for prostate cancer: prostate-specific antigen and beyond. Clin Chem Lab Med. 2020 Feb 25;58(3):326-339. doi: 10.1515/cclm-2019-0693. PMID 31714881
- [Background] Mazzone E, Stabile A, Pellegrino F, Basile G, Cignoli D, Cirulli GO, Sorce G, Barletta F, Scuderi S, Bravi CA, Cucchiara V, Fossati N, Gandaglia G, Montorsi F, Briganti A. Positive Predictive Value of Prostate Imaging Reporting and Data System Version 2 for the Detection of Clinically Significant Prostate Cancer: A Systematic Review and Meta-analysis. Eur Urol Oncol. 2021 Oct;4(5):697-713. doi: 10.1016/j.euo.2020.12.004. Epub 2020 Dec 25. PMID 33358543
- [Background] Sathianathen NJ, Omer A, Harriss E, Davies L, Kasivisvanathan V, Punwani S, Moore CM, Kastner C, Barrett T, Van Den Bergh RC, Eddy BA, Gleeson F, Macpherson R, Bryant RJ, Catto JWF, Murphy DG, Hamdy FC, Ahmed HU, Lamb AD. Negative Predictive Value of Multiparametric Magnetic Resonance Imaging in the Detection of Clinically Significant Prostate Cancer in the Prostate Imaging Reporting and Data System Era: A Systematic Review and Meta-analysis. Eur Urol. 2020 Sep;78(3):402-414. doi: 10.1016/j.eururo.2020.03.048. Epub 2020 May 20. PMID 32444265
- [Background] Berry B, Parry MG, Sujenthiran A, Nossiter J, Cowling TE, Aggarwal A, Cathcart P, Payne H, van der Meulen J, Clarke N. Comparison of complications after transrectal and transperineal prostate biopsy: a national population-based study. BJU Int. 2020 Jul;126(1):97-103. doi: 10.1111/bju.15039. Epub 2020 Apr 6. PMID 32124525
- [Background] Hubner N, Shariat S, Remzi M. Prostate biopsy: guidelines and evidence. Curr Opin Urol. 2018 Jul;28(4):354-359. doi: 10.1097/MOU.0000000000000510. PMID 29847523
- [Background] Tao T, Wang C, Liu W, Yuan L, Ge Q, Zhang L, He B, Wang L, Wang L, Xiang C, Wang H, Chen S, Xiao J. Construction and Validation of a Clinical Predictive Nomogram for Improving the Cancer Detection of Prostate Naive Biopsy Based on Chinese Multicenter Clinical Data. Front Oncol. 2022 Jan 21;11:811866. doi: 10.3389/fonc.2021.811866. eCollection 2021. PMID 35127526
- [Result] Rebello RJ, Oing C, Knudsen KE, Loeb S, Johnson DC, Reiter RE, Gillessen S, Van der Kwast T, Bristow RG. Prostate cancer. Nat Rev Dis Primers. 2021 Feb 4;7(1):9. doi: 10.1038/s41572-020-00243-0. PMID 33542230
- [Result] Naji L, Randhawa H, Sohani Z, Dennis B, Lautenbach D, Kavanagh O, Bawor M, Banfield L, Profetto J. Digital Rectal Examination for Prostate Cancer Screening in Primary Care: A Systematic Review and Meta-Analysis. Ann Fam Med. 2018 Mar;16(2):149-154. doi: 10.1370/afm.2205. PMID 29531107